CLINICAL TRIAL: NCT00719901
Title: A Phase I/II Trial of Obatoclax Mesylate (GX15-070MS) in Combination With Bortezomib for the Treatment of Relapsed Multiple Myeloma
Brief Title: Obatoclax and Bortezomib in Treating Patients With Relapsed or Refractory Multiple Myeloma
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: This trial was terminated due to slow accrual and the drug supply of Obatoclax during the phase I; therefore, the phase II portion will never open.
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2009-00255; NCI-2009-00255 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); CDR0000597950; MAYO-MC068A; MC068A (Other: Mayo Clinic); 7952 (Other: CTEP); N01CM62205 (NIH); P01CA136447 (Other Grant/Funding Number: US NIH Grant/Contract Award Number); N01CM62208 (NIH); N01CM62203 (NIH); NCT01647048 (obsolete NCT alias)
Record Dates: First submitted 2008-07-19; First posted 2008-07-22 (Estimated); Results first posted 2013-12-09 (Estimated); Last update posted 2015-01-12 (Estimated); Status verified 2013-10

CONDITIONS: Refractory Multiple Myeloma; Stage I Multiple Myeloma; Stage II Multiple Myeloma; Stage III Multiple Myeloma
MeSH Terms: conditions — Multiple Myeloma | interventions — obatoclax; Bortezomib

ARMS (1):
- Treatment (enzyme inhibitor therapy) (Experimental): Patients receive obatoclax mesylate IV over 3 hours and bortezomib IV on days 1, 4, 8, and 11. Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: obatoclax mesylate; Drug: bortezomib; Other: laboratory biomarker analysis

INTERVENTIONS:
Drug: obatoclax mesylate — Given IV
  Other Names: GX15-070MS
Drug: bortezomib — Given IV
  Other Names: LDP 341; MLN341; VELCADE
Other: laboratory biomarker analysis — Correlative studies

SUMMARY:
This phase I/II trial is studying the side effects and best dose of obatoclax when given together with bortezomib and to see how well they work in treating patients with relapsed or refractory multiple myeloma. Obatoclax and bortezomib may stop the growth of cancer cells by blocking some of the enzymes needed for cell growth. Giving obatoclax together with bortezomib may kill more cancer cells.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the maximum tolerated dose and recommended phase II dose of obatoclax mesylate when given in combination with bortezomib in patients with relapsed or refractory multiple myeloma. (Phase I) II. To evaluate the response rate (complete response, partial response, and very good partial response) in patients treated with this regimen. (Phase II)

SECONDARY OBJECTIVES:

I. To determine the duration of progression-free and overall survival of these patients.

II. To evaluate the incidence of toxicities of this regimen in these patients. III. To explore the utility of genetic markers based on initial evidence that they are predictive of drug responsiveness and/or successful target inhibition.

OUTLINE: This is a multicenter, phase I, dose-escalation study of obatoclax mesylate followed by a phase II study.

Patients receive obatoclax mesylate IV over 3 hours and bortezomib IV on days 1, 4, 8, and 11. Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed every 3 months until disease progression and then every 6 months for up to 3 years.

ELIGIBILITY:
Inclusion Criteria:

* Symptomatic multiple myeloma, meeting the following criteria at original diagnosis:

  * Bone marrow plasmacytosis with ≥ 10% plasma cells or sheets of plasma cells or biopsy proven plasmacytoma
  * Symptomatic disease (e.g.,anemia, hypercalcemia, bone disease, or renal dysfunction) that requires the initiation of therapy
* Measurable diseases assessed by one of the following:

  * Monoclonal plasma cells detectable in the bone marrow
  * Monoclonal serum spike detectable by serum protein electrophoresis or immunofixation
  * Monoclonal protein detectable in the urine by electrophoresis or immunofixation
  * Abnormal levels of the serum free light chains with an abnormal ratio between kappa and lambda
* Progressive disease after ≥ 1 prior therapy for myeloma
* Previously treated with ≤ 10 courses (30 weeks) of bortezomib and had no disease progression during therapy OR completed bortezomib therapy within the past 6 weeks

  * No prior discontinuation of bortezomib therapy due to drug intolerance
* No known brain metastases
* No intracranial edema, intracranial metastasis, or active epidural disease

  * Patients with lytic lesions of the cranium secondary to myeloma are eligible
* ECOG performance status 0-2
* Life expectancy > 6 months
* ANC ≥ 1,000/mm³
* Platelet count ≥ 50,000/mm³
* Bilirubin normal
* AST and ALT ≤ 2.5 times upper limit of normal (ULN)
* Creatinine ≤ 2 times ULN
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* No peripheral neuropathy > NCI toxicity grade 2
* No history of allergic reactions attributed to compounds of similar chemical or biologic composition to obatoclax mesylate or bortezomib
* No concurrent uncontrolled illness including, but not limited to the following:

  * Ongoing or active infection
  * Symptomatic congestive heart failure
  * Unstable angina pectoris
  * Cardiac arrhythmia, including QTc > 450 msec
  * Psychiatric illness/social situations that would limit compliance with study requirements
* No history of seizure disorder
* No other neurological disorder or dysfunction that, in the opinion of the investigator, would confound the evaluation of neurologic and other adverse events associated with obatoclax mesylate
* At least 14 days since prior chemotherapy and recovered
* More than 28 days since prior experimental drugs and/or investigational agents
* No concurrent CYP interactive medications
* No concurrent combination antiretroviral therapy for HIV-positive patients
* No other concurrent anticancer therapy

  * Growth factors and bisphosphonates are allowed as medically indicated
  * Prednisone (≤ 10 mg per day) allowed provided there has been no dose increase within the past 2 weeks
* No other concurrent investigational agents

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2008-07; Primary Completion 2011-04 (Actual); Study Completion 2012-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alexander Stewart, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from 5 medical clinics in the United States between February 2008 and January 2011.
Pre-assignment Details: This was a phase I/II trial. A total of 11 participants were accrued, all to the phase I portion. This trial was terminated due to slow accrual and the drug supply of Obatoclax during the phase I; therefore, the phase II portion will never open. No results from the phase II portion are available.
Groups:
- Treatment (Enzyme Inhibitor Therapy): Patients receive obatoclax mesylate IV over 3 hours and bortezomib (1.3 mg/m^2) IV on days 1, 4, 8, and 11. Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity.
Period: Overall Study
Arm/Group | Treatment (Enzyme Inhibitor Therapy)
Started | 11
Completed | 0
Not Completed | 11
Not completed — Adverse Event | 5
Not completed — Withdrawal by Subject | 1
Not completed — Alternate Treatment | 1
Not completed — Disease Progression | 3
Not completed — Availability of Study Drug | 1

BASELINE CHARACTERISTICS:
Population: One patient withdrew prior to beginning treatment and was replaced, thus, will be excluded in all analysis.
Arm/Group | Treatment (Enzyme Inhibitor Therapy)
Number analyzed (Participants) | 10
Age, Continuous [Mean (Standard Deviation); unit: years] | 62.1 (10.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 6
Region of Enrollment [Number; unit: participants]
  United States | 10
Performance Status [Number; unit: participants]
  0=Fully active | 1
  1=Restricted in physically strenuous activity | 9
Dose Level [Number; unit: participants]
  Obatoclax mesylate IV 14 mg/m^2 | 3
  Obatoclax mesylate IV 30 mg/m^2 | 4
  Obatoclax mesylate IV 40 mg/m^2 | 3

OUTCOME MEASURES:

1. Primary Outcome: Number of Dose-limiting Toxicity (DLT) Incidents (Phase I)
Description: DLT was defined as any events that is determined to be possibly, probably, or definitely related to the combination of bortezomib and GX15-070 (as determined by the investigator) and occurring during the first cycle of treatment, irrespective of whether the toxicity resolved. Hematologic DLT measures were assessed using the continuous variables as the outcome measures (primarily nadir and percent change from baseline values) as well as categorization via Common Terminology Criteria for Adverse Events (CTCAE) version 3 standard toxicity grading.
Time Frame: Up to 21 days of every first course
Measure: Number; unit: Toxicity Incidents
Arm/Group | Treatment (Enzyme Inhibitor Therapy)
Number analyzed (Participants) | 10
Toxicity Incidents | 4

2. Primary Outcome: Proportion of Patients Who Achieve a Partial Response or Better. (Phase II)
Description: In order to be classified as a hematologic response, confirmation of serum monoclonal protein, serum immunoglobulin free light chain (when primary determinant of response) and urine monoclonal protein (when primary determinant of response) results must be made by verification on two consecutive determinations.
Time Frame: From baseline to up to 3 years
Population: No participants proceeded to Phase II for evaluation.
Arm/Group | Treatment (Enzyme Inhibitor Therapy)
Number analyzed (Participants) | 0

3. Secondary Outcome: Number of Patients Who Have at Least a Partial Response (Phase I)
Description: as for outcome 2
Time Frame: From baseline to up to 3 years
Measure: Number; unit: participants
Arm/Group | Treatment (Enzyme Inhibitor Therapy)
Number analyzed (Participants) | 10
participants | 4

4. Secondary Outcome: Time to Progression (Phase II)
Description: The distribution of time to progression will be estimated using the method of Kaplan-Meier.
Time Frame: Time from registration to the time of progression
Population: No participants proceeded to Phase II for evaluation.
Arm/Group | Treatment (Enzyme Inhibitor Therapy)
Number analyzed (Participants) | 0

5. Secondary Outcome: Overall Survival (Phase II)
Description: The distribution of overall survival will be estimated using the method of Kaplan-Meier.
Time Frame: Time from registration to death due to any cause
Population: No participants proceeded to Phase II for evaluation.
Arm/Group | Treatment (Enzyme Inhibitor Therapy)
Number analyzed (Participants) | 0

6. Secondary Outcome: Time to Treatment Failure (Phase II)
Description: Time to treatment failure will be evaluated using the method of Kaplan-Meier.
Time Frame: Time from study entry to the date patients end treatment
Population: No participants proceeded to Phase II for evaluation.
Arm/Group | Treatment (Enzyme Inhibitor Therapy)
Number analyzed (Participants) | 0

7. Secondary Outcome: Toxicity as Assessed by the National Cancer Institute (NCI) CTCAE v 3.0 (Phase II)
Description: Toxicity is defined as adverse events that are classified as either possibly, probably, or definitely related to study treatment. The maximum grade for each type of toxicity will be recorded for each patient, and frequency tables will be reviewed to determine toxicity patterns. In addition, we will review all toxicities data that is graded as 3, 4, or 5 and classified as either "unrelated or unlikely to be related" to study treatment in the event of an actual relationship developing. Adverse events and toxicities will be evaluated using all patients who have received any study treatment.
Time Frame: From baseline to up to 3 years
Population: No participants proceeded to Phase II for evaluation.
Arm/Group | Treatment (Enzyme Inhibitor Therapy)
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Arm/Group | Treatment (Enzyme Inhibitor Therapy)
Serious Adverse Events (participants affected / at risk) | 3/10
Other Adverse Events (participants affected / at risk) | 10/10
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (Enzyme Inhibitor Therapy) (N=10)
Neutrophil count decreased (Investigations) | 2 (2)
Depressed level of consciousness (Nervous system disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (Enzyme Inhibitor Therapy) (N=10)
Hemoglobin decreased (Blood and lymphatic system disorders) | 10 (36)
Cardiac disorder (Cardiac disorders) | 1 (1)
Diplopia (Eye disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 2 (2)
Diarrhea (Gastrointestinal disorders) | 7 (12)
Nausea (Gastrointestinal disorders) | 4 (7)
Vomiting (Gastrointestinal disorders) | 2 (3)
Fatigue (General disorders) | 5 (6)
Hypersensitivity (Immune system disorders) | 1 (1)
Leukocyte count decreased (Investigations) | 9 (27)
Lymphocyte count decreased (Investigations) | 4 (4)
Neutrophil count decreased (Investigations) | 8 (26)
Platelet count decreased (Investigations) | 8 (23)
Anorexia (Metabolism and nutrition disorders) | 2 (2)
Myalgia (Musculoskeletal and connective tissue disorders) | 4 (10)
Ataxia (Nervous system disorders) | 1 (1)
Depressed level of consciousness (Nervous system disorders) | 1 (1)
Dizziness (Nervous system disorders) | 1 (1)
Extrapyramidal disorder (Nervous system disorders) | 1 (1)
Headache (Nervous system disorders) | 6 (9)
Peripheral motor neuropathy (Nervous system disorders) | 2 (6)
Peripheral sensory neuropathy (Nervous system disorders) | 7 (27)
Speech disorder (Nervous system disorders) | 1 (1)
Anxiety (Psychiatric disorders) | 2 (4)
Depression (Psychiatric disorders) | 1 (2)
Euphoria (Psychiatric disorders) | 4 (6)
Psychosis (Psychiatric disorders) | 3 (3)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 8 (15)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Rash desquamating (Skin and subcutaneous tissue disorders) | 2 (2)

LIMITATIONS AND CAVEATS:
This trial was terminated due to slow accrual and the drug supply of Obatoclax during the phase I; therefore, the phase II portion will never open. No results from the phase II portion are available.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less